CLINICAL TRIAL: NCT02344966
Title: Cohort Study of New Prognostic Factors With Peripheral Blood and Bone Marrow Evaluation at the Time of Diagnosis and During Treatment or Thereafter in Acute Leukemia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2010-0732
Record Dates: First submitted 2014-12-30; First posted 2015-01-26 (Estimated); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Acute Leukemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this study is to evaluate the prognostic factors of acute leukemia patients and to invent the molecular genetic test for sensitive detection of minimal residual disease, and thereby this study would contribute to plan the risk adapted treatment. Patients will have samples of blood and/or bone marrow collected during diagnosis process, treatment and/or thereafter

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with acute leukemia in Severance Hospital.
* Both genders of 16 Years and older
* sign a written informed consent document

Exclusion Criteria:

* No comprehension or willingness to sign a written informed consent document.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Sampling is performed in patients diagnosed with acute leukemia in Severance Hospital.
  Every eligible patients in peroid of study are enrolled. Patients must have the ability and willingness to sign a written informed consent document. Planned number of patients is 1100 considering annual incidence rate.
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2011-06; Primary Completion 2021-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 10years
  Overall survival (OS) is defined as the time from date of diagnosis until death due to any cause within the follow-up period. Surviving patients are censored at date of last contact.

SECONDARY OUTCOMES:
Progression-free survival | 10years
  Progression-free survival (PFS) is defined as survival without disease progression or relapse; patients alive without disease progression or relapse are censored on the last assessment date. Median OS and PFS are calculated using Kaplan-Meier estimates with a 95% confidence interval.
Treatment-related mortality | 10years
  Treatment-related mortality was defined as death unrelated to refractory or progressive disease occurring before first remission was achieved, or any death in complete remission
Complete remission rate | 10 years
  Response assessment is performed according to the criteria reported by BD Cheson et al. (Revised recommendations of the international working group for diagnosis, standardization of response criteria, treatment outcomes, and reporting standards for therapeutic trials in acute myeloid leukemia)

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University College of Medicine, Seoul, South Korea